CLINICAL TRIAL: NCT04620785
Title: PHOTODYNAMIC THERAPY USING METHYLENE BLUE AND INTENSE PULSED LIGHT VERSUS INTENSE PULSED LIGHT ALONE IN TREATMENT OF VERRUCA :A RANDOMIZED CONTROLLED STUDY
Brief Title: Photodynamic Therapy in Treatment of Verrucae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, lecturer of dermatology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0106171
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Verruca Vulgaris
MeSH Terms: conditions — Warts | interventions — Methylene Blue; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- methylene blue/IPL (Experimental): will undergo photodynamic therapy using intralesional 4%methylene blue solution ,after a period of 15 minutes the patient will be subjected to IPL session.
  This will be repeated biweekly until complete clearance of the lesion or a maximum four sessions.
  Interventions: Other: methylene blue / IPL
- IPL (Experimental): will undergo biweekly IPL sessions only until complete clearance of the lesion or a maximum four sessions.
  Interventions: Other: IPL
- saline (Placebo Comparator): will undergo intralesional saline.
  Interventions: Other: saline

INTERVENTIONS:
Other: methylene blue / IPL — therapeutic
  Arms: methylene blue/IPL
Other: IPL — therapeutic
  Arms: IPL
Other: saline — placebo
  Arms: saline

SUMMARY:
To assess the efficacy (clinically and dermoscopically) and safety of photodynamic therapy using intralesional injection of 4% methylene blue solution as a photosensitizer with IPL versus IPL only in treatment of warts.

DETAILED DESCRIPTION:
This study will be conducted on:

Eighty patients suffering of verruca (male and female) divided randomly into three groups: group A, B&C :

Group A: 30 patients will undergo photodynamic therapy using intralesional 4%methylene blue solution and IPL.

Group B: 30 patients will undergo IPL only. Group C (control group):20 patients will undergo intralesional saline.

ELIGIBILITY:
Inclusion Criteria:

1. Age:Above 16 years old.
2. Sex:Both males and female patients.
3. Clinically and dermoscopically documented verruca.
4. No verruca treatment in the last 2 weeks.

Exclusion Criteria:

1. History of photosensitivity disorder.
2. Pregnant and lactating females.
3. Diseases with risk of koebnerization e.g. Psoriasis and Lichen planus.
4. Anogenital warts.
5. Warts on head and neck.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
disappearance of verruca | 10 weeks
  clinical and dermoscopic cure

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided